CLINICAL TRIAL: NCT02253277
Title: A Phase Ib Single-arm, Open-label, Multicenter Study to Assess the Safety and Tolerability of Combined Treatment With Nilotinib 300mg BID and Ruxolitinib Increasing Dose in CML and Ph+ ALL Patients
Brief Title: Safety and Tolerability of Combined Treatment With Nilotinib and Ruxolitinib in CML and Ph+ ALL Patients
Acronym: CoRNea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107YDE19
Record Dates: First submitted 2014-09-17; First posted 2014-10-01 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Chronic Myeloid Leukemia
Keywords: CML, Ph+ ALL
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nilotinib and Ruxolitinib (Experimental): The study included two strata, which were to be treated in parallel. The first stratum consisted of CML-patients in CP, which had been on nilotinib treatment before entering the study. These patients did not optimally respond to the previous treatment. The second stratum consisted of patients with CML in AP or BC and patients with relapsed/refractory Ph+ ALL and Ph+ ALL patients with MRD, with or without previous nilotinib treatment. Patients were treated with 300mg nilotinib BID during the escalation phase (12 months) with increasing doses of ruxolitinib. The dose expansion phase (12 months) began following the determination of the MTD of the combination and the decision to explore the cohort for confirmation of RPIID. In this phase, safety and tolerability of the MTD and/or potential RPIID was to be further evaluated, with the purpose of establishing that this dose is suitable for use in this patient group.
  Interventions: Drug: Nilotinib; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib was supplied by Novartis as 150 mg and 200 mg hard gelatin capsules. Nilotinib was not dosed by weight or body surface area. Medication labels were in German and complied with the legal requirements of Germany. They included storage conditions for the drug but no information about the patient. The investigator emphasized compliance and instructed the patient to take nilotinib exactly as prescribed.
Drug: Ruxolitinib — Ruxolitinib was supplied by Novartis as 5 mg, 15 mg, and 20 mg tablets. Medication labels were in German and complied with the legal requirements of Germany. They included storage conditions for the drug but no information about the patient. The investigator emphasized compliance and instructed the patient to take ruxolitinib exactly as prescribed.

SUMMARY:
In this study it was the rationale to evaluate the safety and tolerability of the combined administration of nilotinib and increasing dose of ruxolitinib in patients with chronic myeloid leukemia and patients with Philadelphia positive acute lymphoblastic leukemia.

ELIGIBILITY:
Inclusion Criteria:

Patients of the first stratum must have chronic myeloid leukemia receiving nilotinib first-line therapy or receiving second-line or subsequent-line treatment with nilotinib.

Patients of the second stratum must have CML in AP/BC or relapsed/refractory Ph+ ALL, or be Ph+ ALL patients with MRD with or without prior nilotinib pretreatment;

Patients must have adequate end organ function, as defined by:

* Creatinine < 2.0 x upper limit of normal (ULN)
* Total bilirubin < 1.5 x ULN (< 3.0 x ULN if related to disease or polymorphism, such as Mb. Gilbert)
* ALT and AST < 2.5 x ULN (< 5.0 x ULN if related to disease)
* Serum lipase ≤ 1.5 x ULN
* Alkaline phosphatase ≤ 2.5 x ULN (< 5.0 x ULN if related to disease);

Patients must have the following electrolyte values within normal limits or corrected to within normal limits with supplements prior to the first dose of study medication:

* Potassium
* Magnesium
* Phosphate
* Total calcium (corrected for serum albumin);

Female patients of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days before initiation of study drug. All WOCBP must use highly effective contraceptive methods throughout and during 3 months after study;

Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1 for patients in CP, ≤ 2 for patients in AP/BC or with relapsed/refractory Ph+ ALL or with Ph+ ALL with MRD;

Patient has the following laboratory values within 7 days of starting study drug:

- For CML and Ph+ ALL patients: platelet count > 75 x 109/L and ANC > 1.0 x 109/L

Exclusion Criteria:

Patient must not have evidence of active malignancy other than the existing CML or ALL

Patient must not receive drugs that interfere with coagulation or inhibits platelet function, with the exception of aspirin ≤ 150 mg per day or low molecular weight heparin.

Patient must not have history of platelet dysfunction, bleeding diathesis, and/or coagulopathy in the 6 months prior to screening;

Patient must not require treatment with any strong CYP3A4 inducer or inhibitor

Patient must not have history of hypersensitivity to any of the study drugs or to drugs of similar chemical classes and their excipients;

Patients must not take other investigational drugs within 28 days prior to screening;

Patient must not be pregnant or lactating at screening and/or baseline;

Patient must not have impaired cardiac functions

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-02-18 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicities (DLTs) | Baseline, up to day 28 (equals first cycle)
  Occurrence of DLTs during cycle 1

SECONDARY OUTCOMES:
Safety and tolerability profile of nilotinib and ruxolitinib administered in combination | Baseline, up to month 12
  Maximum Tolerated Dose (MTD) and/or Recommended Phase II Dose (RPIID) of ruxolitinib in combination with nilotinib. (timeframe, baseline up to month 12)
Trough levels of nilotinib and ruxolitinib administered in combination | Baseline, up to month 12
  Trough levels will be determined by measuring the minimum plasma concentration (Cmin).
Clinical activity of nilotinib and ruxolitinib administered in combination | Baseline and at 3, 6, and 12 months
  Chronic myeloid leukemia in chronic phase: assessment of molecular response: MMR (≤0.1% BCR-ABL) and MR4 (≤0.001% BCR-ABL) at 3, 6, 12 months; Advanced disease: assessment of cytogenetic response will be based on evaluating percentage of Ph+ metaphases

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hochhaus, Prof. Dr. med., Principal Investigator — Jena University Hospital
Locations (4):
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Leipzig

IPD SHARING:
Plan to Share IPD: No